CLINICAL TRIAL: NCT05596864
Title: Application Value of Transabdominal Gastric Contrast Ultrasound in the Diagnosis and Staging Evaluation of Gastric Cancer
Brief Title: Transabdominal Gastric Contrast Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: CUS-GC
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Transabdominal Gastric Contrast Ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Patients with gastric cancer underwent contrast-enhanced CT scan and gastric filling ultrasound, respectively.
  Interventions: Diagnostic Test: gastric contrast ultrasound

INTERVENTIONS:
Diagnostic Test: gastric contrast ultrasound — Gastric contrast ultrasound (GCUS) refers to that the patient fills the stomach cavity with oral water, contrast agent and ultrasound contrast agent before the examination to remove the gas in the stomach cavity and fill the stomach cavity to become a homogeneous echo area and form a good acoustic sound. Interface contrast, more clearly showing the gastric wall hierarchy and the ultrasound examination method of the lesions.
  In this way, not only the changes of the gastrointestinal mucosa can be found, but also the submucosal tumors of the gastrointestinal tract can be clearly displayed, the internal structural characteristics of the tumor, the extent of the lesions, the depth of infiltration, the TNM staging of the tumor, and the lesions of the surrounding organs can be displayed.

SUMMARY:
In this study, the clinical data of patients diagnosed with gastric cancer who were ready for surgery were examined by contrast-enhanced ultrasonography and gastric-enhanced CT before surgery. Based on the results of postoperative pathological examinations, the diagnostic accuracy of gastric filling contrast-enhanced ultrasonography and gastric contrast-enhanced CT in different stages of gastric cancer was compared and analyzed. Provide better guidance for follow-up clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~80 years old, male or female;
2. Diagnosed with gastric cancer by histology or cytology;
3. No distant multiple metastasis;
4. ECOG score 0-2;
5. Heart, lung, liver and kidney function can tolerate surgery;
6. Patients and their families can understand and be willing to participate in this clinical study, and sign the informed consent.

Exclusion Criteria:

1. Previous history of malignant tumor or recent diagnosis combined with other malignant tumors;
2. Patients with gastrointestinal perforation, gastrointestinal bleeding, etc. requiring emergency surgery;
3. Patients with previous gastroduodenal surgery;
4. Preoperative neoadjuvant therapy;
5. Patients and their families refuse surgical treatment;
6. ASA grade ≥ IV and/or ECOG performance status score > 2;
7. Patients with severe liver and kidney function, cardiopulmonary function, coagulation dysfunction or combined with serious underlying diseases who cannot tolerate surgery;
8. Have a history of serious mental illness;
9. Pregnant or lactating women;
10. Patients with other clinical and laboratory conditions considered by the researchers should not participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer who are ready for surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy of gastric contrast ultrasound in judging gastric cancer staging. | one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wei Li, Prof., Principal Investigator — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No